CLINICAL TRIAL: NCT03539796
Title: Dural Puncture Epidural Technique vs. Standard Epidurals vs. Combined-Spinal Epidurals for Cesarean Sections: Does it Really Matter to the Patient?
Brief Title: Epidural Technique: Does it Really Matter to the Patient?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated early because of shortage of supplies with no foreseeable future of when they will be back in stock.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Dawn Manning-Williams, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00098730
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia
Keywords: dural puncture epidurals; DPE; combined-spinal epidural; CSE; cesarean section; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dural puncture epidurals (DPE) (Experimental): Dural puncture epidurals for cesarean section.
  Interventions: Procedure: Dural puncture epidurals (DPE)
- Traditional epidurals (EPI) (Active Comparator): Traditional epidurals (EPI) for cesarean section.
  Interventions: Procedure: Traditional epidurals (EPI)
- Combined-spinal epidural technique (CSE) (Active Comparator): Combined-spinal epidural technique (CSE) for cesarean section.
  Interventions: Procedure: Combined-spinal epidural technique (CSE)

INTERVENTIONS:
Procedure: Dural puncture epidurals (DPE) — Using the Arrow Epidural Kit (AK-05560) an epidural will be placed using the LOR to saline or air technique. A 26g Gertie Marx needle will be inserted through the Touhy epidural needle and used to puncture the dura; clear, free flowing CSF will return in the needle, but no medications will be injected. The 26g spinal needle will be removed, and the epidural catheter inserted through the epidural needle 3-5cm in the epidural space. A test dose with 3mL 1.5% Lidocaine with 1:200,000 epinephrine will be used to confirm the absence of intrathecal or intravascular catheter placement. The epidural catheter will then be dosed with 0.5% Bupivacaine in 5mL increments until a T4 dermatome level is reached. Epidural fentanyl 100mcg will be administered during initial dosing, and morphine-PF 3mg will be given via epidural after delivery of the fetus.
  Arms: Dural puncture epidurals (DPE)
Procedure: Traditional epidurals (EPI) — Using the Arrow Epidural Kit (AK-05560) an epidural will be placed using the LOR to saline or air technique. The catheter will be inserted 3-5cm in the epidural space. A test dose with 3mL 1.5% Lidocaine with 1:200,000 epinephrine will be used to confirm the absence of intrathecal or intravascular catheter placement. The epidural catheter will then be dosed with 0.5% Bupivacaine in 5mL increments until a T4 dermatome level is reached. Epidural fentanyl 100mcg will be administered during initial dosing, and morphine-preservative free (PF) 3mg will be given via epidural after delivery of the fetus.
  Arms: Traditional epidurals (EPI)
Procedure: Combined-spinal epidural technique (CSE) — Using the Arrow Epidural Kit (AK-05560) an epidural will be placed using the LOR to saline or air technique. A 26g Gertie Marx needle will be inserted through the Touhy epidural needle and used to puncture the dura; clear, free flowing CSF will return in the needle and 12mg bupivacaine, 10mcg fentanyl, 200mcg morphine-PF. The 26g spinal needle will be removed, and the epidural catheter inserted through the epidural needle 3-5cm in the epidural space. No epidural test dose will be given immediately compared to the above procedures secondary to intrathecal injection of local anesthetic with this CSE technique. Only after approximately 1 hour after intrathecal injection will a test dose of 3mL 1.5% Lidocaine with 1:200,000 epinephrine will be used to confirm the absence of intrathecal or intravascular catheter placement. The epidural catheter will then be dosed with 0.5% Bupivacaine for the remainder of the procedure if necessary.
  Arms: Combined-spinal epidural technique (CSE)

SUMMARY:
The main objective of this study will be to determine if the dural puncture epidural (DPE) provides superior analgesia and better patient satisfaction when compared to traditional epidurals for cesarean sections, and to also determine if patient satisfaction in the DPE group is comparable to that of the CSE technique.

DETAILED DESCRIPTION:
There are approximately 4 million child birth deliveries in US hospitals per year, and 1.3million of those births are via cesarean section (c-section). With this type of surgery, obstetric anesthesiology plays an important role. The main objective of this study will be to determine if the dural puncture epidural (DPE) provides superior analgesia and better patient satisfaction when compared to traditional epidurals for cesarean sections, and to also determine if patient satisfaction in the DPE group is comparable to that of the CSE technique.

ELIGIBILITY:
Inclusion Criteria:

* Female parturient at Grady Memorial Hospital must meet one of the following:
* Parturient having a scheduled or elective cesarean section
* Parturient not having primary cesarean-section
* At least 18 years of age
* Subject has signed the informed consent

Exclusion Criteria:

* Parturient who is unable or unwilling to sign the consent form
* Parturient having primary cesarean section
* Parturient with known complex cardiac disease (ex…aortic/mitral stenosis, aortic aneurysms, congenital heart disease with residual defects…etc)
* Parturient with any contraindication to neuraxial anesthesia such as coagulopathy, infection, or patient refusal
* Parturient having a fourth or more cesarean section

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 57 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
Percent of patients with Numeric Pain Rating Score (NPRS)<1 in the DPE vs. EPI group | 1 hour after procedure
  The blinded investigator will visit the patient within 1hour of block placement and ask to select Numeric Pain Rating Score (NPRS) (1-10) during procedure. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). Scores range from 0-10 points, with higher scores indicating greater pain intensity.
Percent of patients with Numeric Pain Rating Score (NPRS) <3 in the DPE vs. EPI group. | 1 hour after procedure
  The blinded investigator will visit the patient 3 hours within 1hour of block placement and ask to select Numeric Pain Rating Score (NPRS) (1-10) during procedure.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). Scores range from 0-10 points, with higher scores indicating greater pain intensity.
Percent of patients with Numeric Pain Rating Score (NPRS)<1 in the DPE vs. CSE group | 1 hour after procedure
  The blinded investigator will visit the patient within 1hour of block placement and ask to select Numeric Pain Rating Score (NPRS) (1-10) during procedure.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). Scores range from 0-10 points, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Percent of patients required rescue analgesia in the DPE vs. EPI group | During labor/delivery (up to 24 hours)
  Additional sedation administered during procedure will be documented.
Percent of patients required rescue analgesia in the DPE vs. CSE group | During labor/delivery (up to 24 hours)
  Additional sedation administered during procedure will be documented. .

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Manning-Williams, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System (CRN), Atlanta, Georgia, United States